CLINICAL TRIAL: NCT05307822
Title: CSD210903: A Study to Determine Subject Puffing Patterns of a Heated Tobacco Product With Four Non-Combusted Cigarette Variants in an Ambulatory Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSD210903
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Smoking; Smoking Behaviors; Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Menthol with HTP device (20020064) (Experimental): Subjects will self-assign to one of three menthol flavor variants of non-combusted cigarette products based on their self-reported flavor usage history.
  Interventions: Other: Non-combusted cigarette variant 42001401; Other: Non-combusted cigarette variant 42001399; Other: Non-combusted cigarette variant 40007386
- Cohort 2: Non-Menthol with HTP device (20020064) (Experimental): Subjects will self-assign to a non-menthol flavor variant of a non-combusted cigarette product based on their self-reported flavor usage history.
  Interventions: Other: Non-combusted cigarette variant 42001402

INTERVENTIONS:
Other: Non-combusted cigarette variant 42001401 — Menthol flavor variant of a non-combusted cigarette (42001401)
  Arms: Cohort 1: Menthol with HTP device (20020064)
Other: Non-combusted cigarette variant 42001399 — Menthol flavor variant of a non-combusted cigarette (42001399)
  Arms: Cohort 1: Menthol with HTP device (20020064)
Other: Non-combusted cigarette variant 40007386 — Menthol flavor variant of a non-combusted cigarette (40007386)
  Arms: Cohort 1: Menthol with HTP device (20020064)
Other: Non-combusted cigarette variant 42001402 — Non-Menthol flavor variant of a non-combusted cigarette (42001402)
  Arms: Cohort 2: Non-Menthol with HTP device (20020064)

SUMMARY:
This is a multi-center, open-label, parallel-cohort-study to evaluate the puffing patterns of healthy adult consumers of tobacco products switching from a usual brand (UB) combustible cigarette (CC) and/or a UB Heated Tobacco Product (HTP) to one of four investigational products (IPs), across two heating modes, over a 28-day ambulatory period.

DETAILED DESCRIPTION:
Potential subjects may complete a pre-screening interview and will complete a Screening Visit to assess their eligibility within 28 days prior to enrollment. Based on meeting eligibility requirements, subjects will be scheduled to return to the clinic to complete Enrollment.

This study will recruit adult smokers of both non-menthol and menthol combustible cigarettes, users of non-menthol and menthol HTPs, and dual users of non-menthol and menthol CCs and HTPs.

To minimize bias, subjects will be assigned to either a non-menthol or menthol HTP IP flavor cohort depending upon self-reported flavor usage history. Subjects who report using non-menthol CC/HTP will be assigned to the single non-menthol HTP IP group, and subjects who report using menthol CC/HTP will be assigned to one of the three menthol HTP IP groups after optionally sampling the three menthol HTP IPs and determining which menthol product they would like to use for the length of the study. Once a particular menthol flavor group has reached full enrollment, that flavor will no longer be available for sampling and selection. Subjects will be instructed not to use UB CC or HTP during the study.

At the Enrollment Visit, subjects will be provided a heating device, HTP IPs for their assigned product, a Product Use and Behavior (PUB) instrument, and an electronic device for use with the PUB instrument. The electronic device will have the PUB application installed for topography data capture and PUB data transmission. Subjects will be trained on using the heating device, connecting the PUB instrument, and using the electronic device for PUB data transmission. Based upon their self-reported UB CC and/or HTP usage, subjects will be given a sufficient amount of the assigned HTP IP.

Subjects will be instructed to use the assigned HTP IP in place of UB CC and HTP, as applicable per the subject's normal product use pattern, during the 28-day study period (including a 14-day IP acclimation period followed by a 14-day product use evaluation period). Subjects will be allowed to use non-CC or non-HTP tobacco/nicotine-containing products (e.g., ENDS products (e-cigarettes), snuff, snus, chewing tobacco, modern oral pouches) according to the subject's normal use pattern. The PUB instrument will collect puffing topography data throughout the product use periods.

At the end of the 14-day acclimation period of the study, subjects will receive a phone call from the clinic to assess IP compliance and to ensure that they are not using UB CC or UB HTP and to document any AEs. During the following evaluation period (Days 15-28), subjects will receive a phone call to remind them of guidelines for using their assigned IP and to document any AEs.

At the conclusion of the 28-day ambulatory period, the subjects will return to the clinic, return the heating device, HTP Accessory USB charger and accessories, all unused HTP IPs, the corresponding PUB instrument and its charger, and the electronic device and its charger. Each subject will complete all End of Study procedures including completing the Product Evaluation Scale (PES) questionnaire, two additional questionnaires to assess overall product liking and intention to use, and then subjects will be discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy male or female adults, ≥ 21 years of age, inclusive, at the time of consent.
3. Positive urine cotinine test at the Screening Visit.
4. CC or HTP is the primary form of tobacco- or nicotine-containing products used within 30 days of the Screening Visit. Subjects may be users of other tobacco- or nicotine-containing products. If the subject is a dual/poly user of tobacco- or /nicotine-containing products then the subject must self-report that a CC or HTP is their primary product.
5. Must have used 5 or more CCs or HTP sticks per day over the last 30 days. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of the Screening Visit), or clinical study participation (prior to 30 days of the Screening Visit) will be allowed at the discretion of the Principal Investigator (PI). Dual users of CCs and HTPs (either 5 CCs or 5 sticks per day or a combination of 5 products per day) will also be allowed into the study.
6. Males must use an acceptable method of birth control from Visit 1 until the end of the study, unless they have had a vasectomy or are abstinent from heterosexual intercourse (as a lifestyle choice, not just for the purpose of study participation), or their female partner is not able to bear children.
7. Females must be willing to use a form of contraception acceptable to the PI from the time of signing informed consent until the end of the study.

   Examples of acceptable means of birth control are, but not limited to:
   1. Surgical sterilization (hysterectomy, bilateral tubal ligation/occlusion, bilateral oophorectomy, bilateral salpingectomy);
   2. Established use of oral, implantable, injectable or transdermal methods of contraception associated with inhibition of ovulation;
   3. Physical barrier method (e.g., condom, diaphragm/sponge/cervical cap) with spermicide;
   4. Non-hormone releasing intrauterine devices (IUD) or hormone-releasing IUDs (e.g., Mirena or Kyleena);
   5. Vasectomized partner;
   6. Abstinence from heterosexual intercourse (as a lifestyle choice, not just for the purpose of study participation); and
   7. Post-menopausal and not on hormone replacement therapy.
8. Must be willing to use the assigned IP and only the assigned flavor as their primary source of nicotine use for the full duration of the 28-day ambulatory period. Use of other non-CC or non-HTP tobacco/nicotine-containing products (e.g., ENDS products (e-cigarettes), snuff, snus, chewing tobacco, modern oral pouches) will be permitted during the ambulatory period.
9. Must have familiarity with modern electronic devices such as an IOS/Android smart phone or tablet computer ("tablet") and be willing to be provided with an electronic device, that allows for both Bluetooth connectivity and internet connectivity. Must be willing to use an application on the electronic device and keep the application active for the length of the study
10. Able to safely perform the required study procedures, as determined by the PI.

Exclusion Criteria:

1. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, or neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study participant unsuitable to participate in this clinical study.
2. History of, presence of, or clinical laboratory test results indicating diabetes.
3. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes.
4. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be allowed at the PI's discretion, pending written approval from the Medical Monitor.
5. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that have been surgically and/or cryogenically removed.
6. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
7. Use of any medication or substance that aids in smoking cessation, including but not limited to: NRT (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to signing the ICF.
8. Participation in another clinical trial within (≤) 30 days prior to signing the ICF. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the ICF in the current study.
9. Females who have a positive pregnancy test, or who are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
10. Subjects ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
11. A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at the Screening Visit or Enrollment Visit.
12. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or a previous attempt within (≤) 30 days prior to signing the ICF.
13. Drinks more than 21 servings of alcoholic beverages per week or has a positive alcohol test result at the Screening Visit or Enrollment Visit.
14. Employed by a tobacco or nicotine manufacturing company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
15. Determined by the PI to be inappropriate for this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Arithmetic Mean | 14 days
  Arithmetic Mean puff duration across the final 14 days of data collection

CONTACTS AND LOCATIONS:
Overall Officials: Gary Dull, PhD, Study Director — RAIS
Locations (7):
- United States (7):
  - Wake Research (MTVCR), Sandy Springs, Georgia
  - AMR Lexington, Lexington, Kentucky
  - Rose Research Center, Charlotte, North Carolina
  - High Point Clinical Trials Center, High Point, North Carolina
  - Rose Research Center, Raleigh, North Carolina
  - Benchmark Research, Fort Worth, Texas
  - Benchmark Research, San Angelo, Texas

IPD SHARING:
Plan to Share IPD: No